CLINICAL TRIAL: NCT07110025
Title: Functional Electrical Stimulation With Core Stabilization Exercises in Children With Spastic Diplegia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelsamed Mahmoud Mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahmed_Msc
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Functional Electrical Stimulation; Cerebral Palsy; Core Stability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- functional electrical stimulation and designed physiotherapy program (Experimental): Children in this group will receive the same training program as control group for 30-minutes in addition to functional electrical stimulation using EV-906 DIGITAL transcutaneous electrical nerve stimulation/EMS neuromuscular stimulator device during core stability exercises for 30-minutes 3 sessions/week for 3 months
  Interventions: Other: designed physical therapy program; Other: core stabilization exercise with neuromuscular electrical stimulation
- designed physiotherapy program (Active Comparator): Children in this group will receive designed physiotherapy program for 1 hour including core stability exercises focusing on correcting pelvic tilting and standing balance. Each child will participate for 1 hour, 3 sessions/week for 3 months
  Interventions: Other: designed physical therapy program

INTERVENTIONS:
Other: designed physical therapy program — a one-hour physical therapy program, focusing on abdominal and back muscle activation and improving balance during standing. The program includes exercises like supine on wedges, prone on wedges, weight shifting, and balance training.
Other: core stabilization exercise with neuromuscular electrical stimulation — The text describes various exercises for children to improve their physical abilities. These exercises include bridging, crab, plank, superhero, wheelbarrow walk, and kneeling on balls. The placement of electrodes on the gluteus maximus and rectus abdominis muscles is determined using anatomical landmarks. The electric current is generated using a biphasic symmetrical waveform with pulse width and intensity, and the stimulus frequency is adjusted to 35 Hz. The neuromuscular electric stimulation mode is used in a Synchronous mode.
  Arms: functional electrical stimulation and designed physiotherapy program

SUMMARY:
This study was done to:

* investigate the combined effect of functional electrical stimulation with core stabilization exercises on pelvic tilting in children with spastic diplegia.
* To investigate the combined effect of functional electrical stimulation with core stabilization exercises on standing balance in children with spastic diplegia.

DETAILED DESCRIPTION:
Spastic diaplegia in children affects motor development and muscle tone. Functional electrical stimulation can improve range of motion, muscle strength, walking speed, and gait. Correcting pelvic position is crucial for treating postural weaknesses. Core stability programs are recommended for spastic cerebral palsy children. Rehabilitation programs should focus on restoring normal pelvic alignment to improve overall balance and functional abilities. This study investigates the effect of functional electrical stimulation on rectus abdominis and gluteus maximus muscles and core stabilization exercises in spastic diplegic cerebral palsy children.

ELIGIBILITY:
Inclusion Criteria:

* Their age will range from 4 to 6 years.
* Their degree of spasticity will range from 1 to 1+, according to the modified Ashworth scale.
* Their motor function will be at level Ⅰ & Ⅱ according to gross motor function classification system.
* Their pelvic tilting angle will be more than 7.6°

Exclusion Criteria:

* Musculoskeletal fixed deformities in lower limbs and spine
* Visual or hearing problems
* Epilepsy
* Botulinum toxin injection or orthopedic surgery within past 6 months or within study period

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of muscle tone | at baseline and after 12 weeks
  The modified Ashworth scale will be used to determine the degree of spasticity of the affected lower limb; the child will be in supine position with head in neutral position, and the examiner will moves the knee of affected side through full range of flexion and extensions the child is instructed to stay relaxed and to avoid resisting or facilitating the joint movement applied by the examiner; children with grades 1 or 1+ will be included
Assessment of gross motor function level | at baseline and after 12 weeks
  The Gross Motor Function Classification System is a clinical classification system with five levels based on functional limitations, the need for handheld mobility devices, and movement quality. It includes children with level I and II and those transported in a manual wheelchair.

SECONDARY OUTCOMES:
Assessment of change of pelvic tilting | at baseline and after 12 weeks
  Pelvic inclinometers and pelvic meter (PALM) are devices designed to assess pelvic tilt. Pelvic inclinometers have adjustable arms for direct contact with bony landmarks, while Pelvic inclinometers and pelvic meter have adjustable arms for contact with the anterior superior iliac spine and posterior superior iliac spine. These devices are typically used in a relaxed standing position, with children with a pelvic tilting angle over 7.6° included.
Assessment of change of balance | at baseline and after 12 weeks
  The Humac Balance System is a combination of a balance board and Humac Balance software, providing a robust assessment tool for static and dynamic balance. It offers various training and measurement routines, including weight-bearing random motions, center of pressure, limits of stability, and roadway measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Cairo, Egypt